CLINICAL TRIAL: NCT07120594
Title: Evaluate the Effectiveness of Buffering Local Anesthetic With Sodium Bicarbonate in Infected and Inflamed Teeth in Children
Brief Title: Evaluate Buffering Local Anesthetic in Inflamed Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TishreenU Pedodontic
Record Dates: First submitted 2025-07-24; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2023-10

CONDITIONS: Inflamed and Infected Primary Molars in Children; Effectiveness of Buffered Local Anesthesia During Dental Extraction
Keywords: Buffered local anesthesia; Sodium bicarbonate; Pain during injection; Pediatric dentistry; Tooth extraction
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Local Anesthetic (Active Comparator): Participants receive the standard local anesthetic solution-lidocaine 2% with epinephrine 1:80,000-for extraction of infected and inflamed primary molars.
  Interventions: Drug: Unbuffered lidocaine 2% with epinephrine 1:80,000
- Buffered Local Anesthetic (Experimental): Participants receive a buffered local anesthetic solution-lidocaine 2% with epinephrine 1:80,000 buffering with sodium bicarbonate-to assess enhanced anesthetic efficacy during extraction of infected and inflamed primary molars.
  Interventions: Drug: Buffered lidocaine 2% with epinephrine 1:80,000

INTERVENTIONS:
Drug: Unbuffered lidocaine 2% with epinephrine 1:80,000 — Standard local anesthetic solution without pH modification. Used for maxillary extraction of infected primary molars in pediatric patients.
  Arms: Standard Local Anesthetic
Drug: Buffered lidocaine 2% with epinephrine 1:80,000 — Local anesthetic solution mixed with sodium bicarbonate to increase pH before injection. Used for maxillary extraction of infected primary molars in pediatric patients.
  Arms: Buffered Local Anesthetic

SUMMARY:
This randomized, double-blinded, split-mouth clinical trial evaluates the effect of buffering local anesthetic with sodium bicarbonate in pediatric dental extractions. Twenty children aged 6 to 10 years with two infected primary molars on opposite sides of the maxilla participated. Each child received standard anesthetic on one side and buffered anesthetic on the other. Pain levels and onset time were measured to assess anesthetic efficacy.

DETAILED DESCRIPTION:
This randomized, controlled, double-blinded, split-mouth clinical trial aims to evaluate the efficacy of buffering local anesthetic solution with sodium bicarbonate in the extraction of infected and inflamed primary molars in children. Infected tissues tend to have a lower PH , which can limit the effectiveness of local anesthetics by reducing the proportion of the active, non-ionized drug form. buffering with sodium bicarbonate improve anesthetic performance by raising the pH of the solution, enhancing its diffusion and clinical effectiveness.

The study included 20 healthy children aged 6 to 10 years, each with two infected or inflamed primary molars located on opposite sides of the maxilla. A split-mouth design was employed, where each child received a standard local anesthetic solution - lidocaine 2% with epinephrine 1:80,000 - on one side, and a buffered solution (alkalinized with sodium bicarbonate) on the contralateral side.

To assess anesthetic efficacy, three parameters were measured: pulse rate (as a physiologic indicator of pain), the Sound-Eye-Motor (SEM) scale (for behavioral response), and the Wong-Baker Faces Pain Rating Scale (for subjective pain reporting). Onset time of anesthesia was also recorded.

The study aims to determine whether buffering lidocaine with sodium bicarbonate improves pain control and onset time during pediatric dental extractions in inflamed and infected tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6 to 10 years with bilateral maxillary first or second primary molars indicated for extraction due to infection and inflammation.
2. Presence of clinical signs of inflammation (e.g., redness, swelling) in the gingiva surrounding the affected teeth.
3. Medically healthy children with no systemic diseases or cognitive disabilities.
4. Children with positive or definitely positive behavior according to the Frankl Behavior Rating Scale.
5. No intake of medications that may interfere with pain perception during the 24 hours preceding the treatment session.

Exclusion Criteria:

1. Presence of systemic medical conditions.
2. Children with negative or definitely negative behavior according to the Frankl Behavior Rating Scale.
3. Known allergy to the local anesthetic agent.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Pain level during tooth extraction in inflamed sites (self-reported) | During the tooth extraction procedure
  Procedural pain during extraction was assessed using the Wong-Baker FACES Pain Rating Scale to measure children's self-reported pain. This scale uses six cartoon faces representing increasing levels of pain, scored from 0 (no pain) to 10 (worst pain). Children were asked to indicate the face that best matched their pain level during tooth extraction in inflamed areas. Higher scores indicate greater pain intensity.
Pain-related behavioral response during extraction in inflamed primary molars (observer-rated) | During the tooth extraction procedure
  Procedural pain behavior will be assessed using the Sound-Eye-Motor (SEM) scale. Trained observers will score behavioral responses during extraction; higher scores indicate stronger pain-related behavior.
Physiological response during extraction in inflamed primary molars (heart rate) | through the extraction procedure
  Heart rate (beats per minute) will be continuously monitored with a pulse oximeter. Increases from baseline are considered indicators of pain/stress during extraction.

SECONDARY OUTCOMES:
Pain perception during injection of anesthetic solution (self-reported) | During and within 1 minute after anesthetic injection
  Pain during injection will be self-reported using the Wong-Baker FACES Pain Rating Scale. Children indicate the face that best matches injection pain (0-10)
Behavioral response during anesthetic injection (SEM) | During and within 1 minute after anesthetic injection
  Observer-rated SEM scores will be recorded during anesthetic injection to evaluate behavioral response to injection pain
Physiological response to injection (heart rate) | During anesthetic injection
  Heart rate (beats per minute) will be recorded before, during, and immediately after injection. Changes from baseline will be used as an objective marker of pain/stress

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dentistry, Tishreen University, Latakia, Latakia Governorate, Syria

IPD SHARING:
Plan to Share IPD: No